CLINICAL TRIAL: NCT00068341
Title: Neoadjuvant Treatment and Molecular Characterization of Locally Advanced Breast Cancer
Brief Title: Docetaxel and Carboplatin With or Without Trastuzumab Before Surgery in Treating Women With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-11-084; CDR0000321924; AVENTIS-GIA-11156; GENENTECH-H2269s
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (neoadjuvant therapy) (Experimental): see intervention description
  Interventions: Drug: carboplatin; Drug: docetaxel; Biological: trastuzumab
- Arm II (neoadjuvant therapy) (Experimental): please see intervention description
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: docetaxel
- HER2/neu negative patients (Experimental): please see intervention description
  Interventions: Drug: carboplatin; Drug: docetaxel

INTERVENTIONS:
Biological: trastuzumab — Cycle 5-7 post-op only Day 1 4mg/kg IV Day 8, 15 2mg/kg IV Cycle 8 Cycle 8 Day 1, 8, 15 2mg/kg IV Day 22 6mg/kg IV
  Other Names: Herceptin
  Arms: Arm II (neoadjuvant therapy)
Drug: carboplatin — Cycle 1-8 Day 1 or 2 AUC = 6 IV
Drug: docetaxel — Cycle 1-8 Day 1 or 2: 75 mg/m2 IV
  Other Names: Taxotere
Biological: trastuzumab — Cycle 1-4 pre-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
  Cycle 5-7 post-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
  Cycle 8 Day 1, 8, 15 2mg/kg IV Day 22 6mg/kg IV
  Other Names: Herceptin
  Arms: Arm I (neoadjuvant therapy)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether docetaxel and carboplatin are more effective with or without trastuzumab in treating breast cancer.

PURPOSE: This randomized phase II trial is studying how well giving docetaxel together with carboplatin and trastuzumab before surgery works compared to docetaxel and carboplatin alone before surgery in treating women with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed infiltrating adenocarcinoma of the breast
* Primary breast cancer > 5cm, or skin/chest wall involvement, any N, without evidence of metastasis.
* No prior radiation to the involved breast
* ECOG (Electrocochleography) performance status 0-2
* Age 18 years to 80 years
* Absolute Neutrophil count > 1500 cell/μl, platelet count > 100000 cells/μl and hemoglobin > 9 g/dl
* All liver function tests < upper limit of normal
* Serum creatinine < 2.0 mg/dl
* Normal left ventricular ejection fraction (LVEF) as determined by MUGA (Multiple Gated Acquisition) scan or echocardiogram
* HER-2/neu status is determined by a FISH (Fluorescence in situ hybridization) test. [FISH (+) is HER-2/neu (+)]
* If female of childbearing potential, pregnancy test is negative
* If premenopausal and not surgically sterilized, the patient agrees to use effective birth control method for the duration of the study
* Informed consent has been obtained

Exclusion Criteria:

* Non-confirmed infiltrating adenocarcinoma breast cancer
* Evidence of metastasis
* Previous chemotherapy using the drugs proposed in this study, specifically Herceptin®, Taxotere®, and/or Carboplatin
* Prior radiation to the involved breast
* Recent breast cancer drug therapy within last 5 years of any form
* History of allergy to polysorbate or castor oil
* Ongoing active infection
* Concurrent life-limiting disease with a life expectancy of less than one year
* Past or current history of other malignancy within the past 5 years which could affect the diagnosis or assessment of breast cancer, except for curatively treated non-melanoma skin cancer and/or in situ carcinoma of the cervix
* Pregnancy, nursing, fertile women who do not use birth control device
* Inability to give informed consent
* Patients with pre-existing peripheral neuropathy > grade 2

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena R. Chang, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Wilshire Oncology Medical Group, Incorporated - Pomona, Pomona, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 2002-2007 Types of location: oncology outpatient clinics
Groups:
- Arm I (Neoadjuvant Therapy): see intervention description
  carboplatin: Cycle 1-8 Day 1 or 2 AUC = 6 IV (AUC = area under the curve, total drug exposure over time)
  docetaxel: Cycle 1-8 Day 1 or 2: 75 mg/m2 IV
  trastuzumab: Cycle 1-4 pre-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
  Cycle 5-7 post-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
  Cycle 8 Day 1, 8, 15 2mg/kg IV Day 22 6mg/kg IV
Period: Overall Study
Arm/Group | Arm I (Neoadjuvant Therapy) | Arm II (Neoadjuvant Therapy) | HER2/Neu Negative Patients
Started | 15 | 15 | 44
Completed | 15 | 15 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Neoadjuvant Therapy): see intervention description
  carboplatin: Cycle 1-8 Day 1 or 2 AUC = 6 IV
  docetaxel: Cycle 1-8 Day 1 or 2: 75 mg/m2 IV
  trastuzumab: Cycle 1-4 pre-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
  Cycle 5-7 post-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
  Cycle 8 Day 1, 8, 15 2mg/kg IV Day 22 6mg/kg IV
- Total: Total of all reporting groups
Arm/Group | Arm I (Neoadjuvant Therapy) | Arm II (Neoadjuvant Therapy) | HER2/Neu Negative Patients | Total
Number analyzed (Participants) | 15 | 15 | 44 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 44 | 74
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 44 | 74
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 44 | 74

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Objective Response Rate of Patients Treated With Taxotere/Carboplatin With or Without Herceptin Preoperatively.
Description: Objective response rate of patients treated with Taxotere/carboplatin with or without Herceptin preoperatively. Objective response equals the combination of complete response (CR), partial response (PR) and marginal response (MR).
  Tumor size was assessed by (1) physical examination, (2) mammography and (3) MRI. 5 response groups: complete response (CR), partial response (PR), marginal response (MR), stable disease (SD) & disease progression (DP). Pathologic response assigned into 2 groups: pCR and non-pCR. pCR-no evidence of residual invasive disease in specimen.
Time Frame: 5 years
Population: pCR was not assessed for 2 patients in the HER2 - (Pre-Op TC) group [1 protocol violation, 1 bilateral disease] and for 1 patient in the HER2+ (Pre-Op TC, Post-Op Herceptin) group [protocol violation]
Measure: Number; unit: participants
Groups:
- Arm I: HER2+: (Pre-Op TCH)
- Arm II: HER2+: (Pre-Op TC, Post-Op Herceptin)
- HER2-: (Pre-Op TC)
Arm/Group | Arm I: HER2+ | Arm II: HER2+ | HER2- | Total
Number analyzed (Participants) | 15 | 14 | 42 | 71
participants
  DFS (Disease Free Survival) | 13 | 8 | 33 | 54
  OS (overall survival) | 13 | 11 | 39 | 63

2. Secondary Outcome: Clinical Tumor Response by Physical Exam and Imaging Studies
Time Frame: 5 years
Population: Clinical response was not assessed for 2 patients in the HER2 - (Pre-Op TC) group [1 protocol violation, 1 bilateral disease] and for 1 patient in the HER2+ (Pre-Op TC, Post-Op Herceptin) group [protocol violation]
Measure: Number; unit: participants
Groups:
- Arm I: Her2+; Arm II:Her2+; Arm III: Her2-: all evaluated subjects.
Arm/Group | Arm I: Her2+ | Arm II:Her2+ | Arm III: Her2-
Number analyzed (Participants) | 15 | 13 | 43
participants
  Complete Response | 8 | 5 | 18
  Partial Response | 7 | 7 | 21
  Marginal Response | 0 | 1 | 4

3. Secondary Outcome: Tumor Response Assessment
Description: Measured by physical examination compared to breast mammography and MRI assessment
Time Frame: 5 years
Population: pCR was not assessed for 2 patients in the HER2 - (Pre-Op TC) group [1 protocol violation, 1 bilateral disease] and for
  1 patient in the HER2+ (Pre-Op TC, Post-Op Herceptin) group [protocol violation]"
Measure: Number; unit: participants
Groups:
- Arm I: Her2 +; Arm II: Her2 +; Arm III: Her -: all enrolled subjects
Arm/Group | Arm I: Her2 + | Arm II: Her2 + | Arm III: Her -
Number analyzed (Participants) | 15 | 13 | 43
participants | 6 | 1 | 12

4. Secondary Outcome: Clinico-histologic Predictors of pCR (Pathologic Complete Response)
Time Frame: 5 years
Population: ER (estrogen-receptor), PR (progesterone-receptor), HER2 (human epidermal growth factor receptor 2), FISH (Fluorescence in situ hybridization), IDC (invasive ductal carcinoma), ILC (invasive lobular carcinoma),
Measure: Number; unit: participants
Groups:
- Pathologic CR - Yes; Pathologic CR - No: All enrolled subjects
Arm/Group | Pathologic CR - Yes | Pathologic CR - No
Number analyzed (Participants) | 74 | 74
participants
  ER-negative | 11 | 14
  ER-positive | 8 | 38
  PR-negative | 14 | 24
  PR-positive | 5 | 28
  ER and PR both negative | 9 | 14
  ER and PR one negative | 7 | 10
  ER and PR both positive | 3 | 28
  HER2 negative | 12 | 30
  HER2 positive | 7 | 22
  T-Stage T2 | 5 | 9
  T-Stage T3 | 13 | 27
  T-Stage T4 | 1 | 16
  Tumor Type - IDC only | 19 | 38
  Tumor Type - all others (compared to IDC only) | 0 | 14
  Tumor Type - ILC only | 0 | 9
  Tumor Type - all other comparted to (ICL only) | 19 | 43
  Triple Negative-yes | 6 | 5
  Triple Negative-no | 7 | 38
  FISH positive Herceptin No | 1 | 13
  FISH positive Herceptin Yes | 6 | 9

5. Secondary Outcome: Pathologic Nodal Status
Description: According to Primary Tumor Response Pathologic lymph node status N0 Axillary and other nearby lymph nodes do not have cancer (when looked at under a microscope) N1 Micrometastases (very small clusters of cancer) OR 1-3 axillary lymph nodes have cancer AND/OR Internal mammary nodes have tiny amounts of cancer found on sentinel node biopsy N2 4-9 axillary lymph nodes have cancer OR Internal mammary nodes have cancer, but axillary lymph nodes do not have cancer N3 10 or more axillary lymph nodes have cancer OR Infraclavicular (under the clavicle) nodes have cancer OR Internal mammary nodes have cancer plus 1 or more axillary lymph nodes have cancer OR 4 or more axillary lymph nodes have cancer plus internal mammary nodes have cancer or micrometastases found on sentinel node biopsy OR Supraclavicular (above the clavicle) nodes have cancer
Time Frame: 5 years
Population: only 71 subjects of the 74 subjects could be analyzed for this outcome measure due to data collection error.
Measure: Number; unit: participants
Groups:
- Arm I (Pre-op TCH); Her2+ (Pre-op TC, Post-op Herceptin); Her2- (Pre-op TC): enrolled subjects
Arm/Group | Arm I (Pre-op TCH) | Her2+ (Pre-op TC, Post-op Herceptin) | Her2- (Pre-op TC)
Number analyzed (Participants) | 15 | 14 | 42
participants
  N(0) | 9 | 4 | 21
  N+ | 6 | 11 | 23

ADVERSE EVENTS:
Time Frame: 3 years from 1st study drug administration
Groups:
- Arm I: HER+ (Pre-Op TCH): Arm I carboplatin: Cycle 1-8 Day 1 or 2 AUC = 6 IV docetaxel: Cycle 1-8 Day 1 or 2: 75 mg/m2 IV trastuzumab: Cycle 1-4 pre-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV
- Arm II: HER2+ (Pre-Op TC, Post-Op Herceptin): Arm II trastuzumab: Cycle 5-7 post-op only Day 1 4mg/kg IV Day 8, 15 2mg/kg IV Cycle 8 Cycle 8 Day 1, 8, 15 2mg/kg IV Day 22 6mg/kg IV carboplatin: Cycle 1-8 Day 1 or 2 AUC = 6 IV docetaxel: Cycle 1-8 Day 1 or 2: 75 mg/m2 IV Cycle 5-7 post-op Day 1 4mg/kg IV Day 8, 15 2mg/kg IV Cycle 8 Day 1, 8, 15 2mg/kg IV Day 22 6mg/kg IV
- Arm III: HER2- (Pre-Op TC): HER2/neu negative patients carboplatin: Cycle 1-8 Day 1 or 2 AUC = 6 IV docetaxel: Cycle 1-8 Day 1 or 2: 75 mg/m2 IV
Arm/Group | Arm I: HER+ (Pre-Op TCH) | Arm II: HER2+ (Pre-Op TC, Post-Op Herceptin) | Arm III: HER2- (Pre-Op TC) | Total
All-Cause Mortality (participants affected / at risk) | 6/15 | 4/14 | 10/45 | 20/74
Serious Adverse Events (participants affected / at risk) | 6/15 | 4/14 | 10/45 | 20/74
Other Adverse Events (participants affected / at risk) | 15/15 | 12/14 | 45/45 | 72/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: HER+ (Pre-Op TCH) (N=15) | Arm II: HER2+ (Pre-Op TC, Post-Op Herceptin) (N=14) | Arm III: HER2- (Pre-Op TC) (N=45) | Total (N=74)
Severe Dehydration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
febrile neutropenia (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 9 (9)
hypokalemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper Extremity Cellulites (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
diarrhea and dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
pain, swelling, mastectomy site cellulitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
death progressive disease (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
divetricular abscess (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: HER+ (Pre-Op TCH) (N=15) | Arm II: HER2+ (Pre-Op TC, Post-Op Herceptin) (N=14) | Arm III: HER2- (Pre-Op TC) (N=45) | Total (N=74)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (14) | 11 (21) | 36 (50) | 59 (85)
Anemia (Blood and lymphatic system disorders) | 13 (42) | 11 (50) | 32 (83) | 56 (175)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3) | 5 (5)
ALT Elevated (Investigations) | 3 (3) | 2 (7) | 8 (13) | 13 (23)
APT Elevated (Investigations) | 2 (2) | 2 (2) | 8 (11) | 12 (15)
AST Elevated (Investigations) | 2 (3) | 3 (3) | 7 (10) | 12 (16)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (3) | 6 (7)
Albumin Decreased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 2 (5) | 13 (47) | 17 (56)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2) | 3 (5)
Appetite Change (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 10 (12) | 16 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 10 (17) | 16 (24)
Blurry Vision (Eye disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Body Ache (Musculoskeletal and connective tissue disorders) | 7 (19) | 11 (23) | 19 (35) | 37 (77)
Chest Complain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 5 (6) | 8 (10)
Chills (General disorders) | 3 (6) | 4 (4) | 2 (2) | 9 (12)
Cold Symptons (General disorders) | 2 (2) | 3 (6) | 7 (13) | 12 (21)
Constipation (Gastrointestinal disorders) | 6 (10) | 5 (7) | 24 (52) | 35 (69)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 1 (1) | 6 (7)
Diarrhea (Metabolism and nutrition disorders) | 5 (19) | 8 (8) | 19 (26) | 32 (53)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2) | 3 (3) | 9 (10)
Dry Mucosa (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (5) | 6 (8)
Edema (General disorders) | 7 (7) | 5 (15) | 3 (3) | 15 (25)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Eye Tearing (Eye disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Fever (General disorders) | 3 (5) | 3 (5) | 1 (1) | 7 (11)
Headache (Nervous system disorders) | 5 (8) | 2 (3) | 13 (16) | 20 (27)
Hot Flashes (Vascular disorders) | 2 (2) | 1 (1) | 8 (8) | 11 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 6 (12) | 8 (14)
Hypersensitivity (General disorders) | 1 (1) | 0 (0) | 6 (8) | 7 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 2 (2) | 5 (7)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 3 (7) | 6 (9) | 13 (20)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 3 (3) | 5 (6)
Indigestion (Gastrointestinal disorders) | 2 (3) | 6 (11) | 12 (17) | 20 (31)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (4) | 4 (7) | 10 (14)
Irregular Menstruation (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 4 (4) | 6 (7)
Leukopenia (Blood and lymphatic system disorders) | 7 (29) | 4 (50) | 17 (116) | 28 (195)
Hot Flashes (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 8 (8) | 11 (11)
Hypergylcemia (Endocrine disorders) | 2 (2) | 0 (0) | 6 (12) | 8 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 2 (2) | 5 (7)
Leukopenia (Blood and lymphatic system disorders) | 13 (29) | 7 (50) | 31 (116) | 51 (195)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7) | 4 (30) | 17 (38) | 28 (75)
Mouth Sore (Gastrointestinal disorders) | 10 (18) | 8 (12) | 11 (21) | 29 (51)
Nail Change (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 11 (12) | 19 (20)
Nausea (Gastrointestinal disorders) | 13 (34) | 12 (45) | 32 (106) | 57 (185)
Neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 10 (25) | 8 (35) | 34 (116) | 52 (176)
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 4 (5) | 6 (8)
Numbness/Tingling (Nervous system disorders) | 6 (8) | 6 (7) | 10 (17) | 22 (32)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (8) | 1 (1) | 9 (11)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (6) | 5 (6) | 12 (15)
Skin Changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Sweats (General disorders) | 2 (4) | 2 (3) | 7 (9) | 11 (16)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Taste Change (General disorders) | 5 (8) | 6 (7) | 15 (20) | 26 (35)
Throat Complaint (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (19) | 8 (24) | 22 (52) | 39 (95)
Vision Change (Eye disorders) | 1 (1) | 0 (0) | 4 (5) | 5 (6)
Vomiting (Gastrointestinal disorders) | 8 (25) | 4 (5) | 16 (30) | 28 (60)
Weakness/Fatigue (General disorders) | 13 (34) | 12 (37) | 41 (155) | 66 (226)
Weight Change (General disorders) | 2 (2) | 0 (0) | 4 (5) | 6 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No